CLINICAL TRIAL: NCT03794297
Title: A Phase II Therapeutic Trial of the Use of Dabrafenib and Trametinib in Patients With BRAF V600 Mutation Positive Lesions in Erdheim Chester Disease
Brief Title: Dabrafenib and Trametinib in Treating Patients With Erdheim Chester Disease With BRAF V600 Mutations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-03659; NCI-2018-03659 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI9598B; 9598B (Other: M D Anderson Cancer Center); 9598B (Other: CTEP); P30CA016672 (NIH)
Record Dates: First submitted 2019-01-01; First posted 2019-01-07 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Erdheim-Chester Disease
MeSH Terms: conditions — Erdheim-Chester Disease | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dabrafenib mesylate, trametinib dimethyl sulfoxide) (Experimental): Patients receive dabrafenib mesylate PO BID and trametinib dimethyl sulfoxide PO QD on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dabrafenib Mesylate; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Drug: Dabrafenib Mesylate — Given PO
  Other Names: Dabrafenib Methanesulfonate; GSK2118436 Methane Sulfonate Salt; GSK2118436B; Tafinlar
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist

SUMMARY:
This phase II trial studies the side effects and how well dabrafenib and trametinib work in treating patients with Erdheim Chester disease that have BRAF V600 gene mutations. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To study the efficacy and safety of dabrafenib mesylate (dabrafenib) and trametinib dimethyl sulfoxide (trametinib) as combination therapy in patients with BRAF V600E positive Erdheim Chester disease.

II. To determine the clinical response rate to dabrafenib and trametinib combination therapy in patients with BRAF V600E positive Erdheim Chester disease.

SECONDARY OBJECTIVES:

I. To determine time response, progression free survival and overall survival. II. To assess disease resistance to this combination therapy.

EXPLORATORY OBJECTIVES:

I. To monitor the degree of histiocytic infiltration-fibrosis progression, stability and regression under combination therapy using fludeoxyglucose F 18 (FDG)-positron emission tomography (PET) scan, magnetic resonance imaging (MRI) scans, computed tomography (CT) scans and technetium (T)-99m bone scans.

II. To monitor serum C-reactive protein (CRP), estrogen receptor (ESR), and cytokine levels as inflammatory markers prior to and during combination therapy.

III. To monitor renal function prior to and during combination therapy in order to assess for functional improvement.

IV. To evaluate the level of functioning, fatigue, motor skills and ability to perform routine daily activities prior to and during therapy in order to assess for improvements in these areas as well as quality of life improvement.

V. To establish duration of treatment-endpoints in patients with BRAF V600E positive Erdheim-Chester disease (ECD) lesions.

OUTLINE:

Patients receive dabrafenib mesylate orally (PO) twice daily (BID) and trametinib dimethyl sulfoxide PO once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients can be previously or simultaneously enrolled in the natural history ECD protocol #11-HG-0207, "Clinical and Basic Investigations into Erdheim Chester disease". Eligible patients must have been diagnosed with Erdheim Chester disease, confirmed by pathological evaluation of the affected tissue with adequate staining. Affected tissue must harbor the BRAF V600 mutation
* Patients must have measurable or evaluable disease according to Response Evaluation Criteria in Solid Tumors 1.1
* Prior treatment, involving interferon, anakinra, imatinib, steroids, chemotherapy with, but not limited to cladribine, vinblastine, 6-mercaptopurine and etoposide, or other medications used empirically for the treatment of ECD, will be acceptable. These therapies should have been completed and discontinued 4 weeks or for biologic agents 4 weeks or 5 half-lives (whichever comes shorter) prior to enrollment in this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)

  * Exception will be made for patients with ECOG performance status =< 3 and Karnofsky performance scale >= 50%, who require the use of wheelchairs, walkers or canes as well as assistance with daily routines secondary to disabilities caused by ECD cerebellar or brain disease that has been stable for >= 3 months
* Life expectancy of greater than 3 months
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Patients must have BRAF V600 mutation in the tumor tissue and/or cell-free deoxyribonucleic acid (DNA), identified by a Clinical Laboratory Improvement Act (CLIA)-certified lab
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 8 g/dL
* Platelets >= 75 x 10^9/L
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) except subjects with known Gilbert's syndrome
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x institutional ULN
* Serum creatinine =< 1.5 x institutional ULN
* Left ventricular ejection fraction >= institutional lower limit of normal (LLN) by echocardiogram (ECHO)
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration or randomization
* Pregnancy and breast feeding. The effects of dabrafenib and trametinib on the developing human fetus are unknown. For this reason women of child-bearing potential must agree to use adequate contraception (barrier method of birth control, or abstinence; hormonal contraception is not allowed due to drug-drug interactions which can render hormonal contraceptives ineffective) for the duration of study participation, and for at least 2 weeks after treatment with dabrafenib or for 4 months after dabrafenib in combination with trametinib. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Based on studies in animals, it is also known that dabrafenib may cause damage to the tissue that makes sperm. This may cause sperm to be abnormal in shape and size and could lead to infertility, which may be irreversible. Safety and efficacy of the combination of dabrafenib and trametinib in pediatric populations have not been investigated. Dabrafenib or trametinib-dabrafenib combination should not be administered to pediatric populations outside clinical trials
* Therapeutic level dosing of warfarin can be used with close monitoring of prothrombin time (PT)/international normalized ratio (INR) by the site. Exposure may be decreased due to enzyme induction when on treatment, thus warfarin dosing may need to be adjusted based upon PT/INR. Consequently, when discontinuing dabrafenib, warfarin exposure may be increased and thus close monitoring via PT/INR and warfarin dose adjustments must be made as clinically appropriate. Prophylactic low dose warfarin may be given to maintain central catheter patency
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Inability to provide informed consent
* Patients treated with prior BRAF and/or MEK inhibitors
* Current use of a prohibited medication. Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A or CYP2C8 are ineligible. Current use of, or intended ongoing treatment with: herbal remedies (e.g., St. John's wort), or strong inhibitors or inducers of P-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1) should also be excluded
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0) grade 2 or higher from previous anti-cancer therapy, except alopecia, at the time of randomization
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dabrafenib
* A history of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (with the exception of cleared HBV and HCV infection, which will be allowed)
* Presence of active malignancy other than the study indication
* Patients with known RAS in ECD, or history of other malignancies with RAS mutations
* Leptomeningeal or brain metastases are allowed. Subjects on a stable dose of corticosteroids can be enrolled with approval of the principal investigator (PI) and Cancer Therapy Evaluation Program (CTEP) medical monitor. Subjects must not receive enzyme-inducing anticonvulsants
* History or evidence of cardiovascular risks, except stable ECD cardiac lesion, including any of the following:

  * QT interval corrected for heart rate using the Bazett's formula (QTcB) >= 480 msec
  * History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within the past 24 weeks prior to randomization
  * History or evidence of current class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Intra-cardiac defibrillators
  * Abnormal cardiac valve morphology (>= grade 2) documented by ECHO; (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study
  * History or evidence of current clinically significant uncontrolled cardiac arrhythmias; clarification: subjects with atrial fibrillation controlled for > 30 days prior to dosing are eligible
  * Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO)
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dabrafenib/trametinib, breastfeeding should be discontinued prior to treatment with dabrafenib/trametinib. These potential risks may also apply to other agents used in this study
* History of retinal vein occlusion (RVO)
* Interstitial lung disease or pneumonitis not secondary to ECD
* Central serous retinopathy (CSR) including presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or visible pathology (e.g., evidence of optic disc cupping, evidence of new visual field defects on automated perimetry, or intraocular pressure > 21 mmHg as measured by tonography) as assessed by ophthalmic examination
* Inability to travel to the treating center
* Patients with confirmed diagnosis of ECD that are asymptomatic and with no visceral involvement are not eligible for this trial (patients with no target lesions as per RECIST 1.1 criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Clinical response rate | Up to 48 weeks after completion of study treatment
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Response to therapy will be evident on follow up imaging studies revealing a decrease in lesion size of 30% or more, which is defined as a partial response as per RECIST criteria, when compared to baseline studies.
Incidence of toxicities | Up to 48 weeks after completion of study treatment
  Assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Time to response | Up to 48 weeks after completion of study treatment
  Will be reported using Kaplan-Meier curves and appropriate 95% confidence intervals.
Duration of response | From the time measurement criteria are met for complete or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 48 weeks after completion of study treatment
  Will be reported using Kaplan-Meier curves and appropriate 95% confidence intervals.
Progression-free survival | From start of treatment to time of progression or death, whichever occurs first, assessed up to 48 weeks after completion of study treatment
  Will be reported using Kaplan-Meier curves and appropriate 95% confidence intervals.
Overall survival | Up to 48 weeks after completion of study treatment
  Will be reported using Kaplan-Meier curves and appropriate 95% confidence intervals.
Degree of histiocytic infiltration using fludeoxyglucose (FDG) positron emission tomography (PET)/computed tomography (CT) and bone scans | Up to 48 weeks after completion of study treatment
Levels of C-reactive protein | Up to 48 weeks after completion of study treatment
Levels of estrogen receptor (ESR) | Up to 48 weeks after completion of study treatment
Levels of cytokines | Up to 48 weeks after completion of study treatment
Change in fatigue | Baseline up to 48 weeks after completion of study treatment
  Patients will be evaluated using the multi-dimensional fatigue inventory.
Change in level of functioning | Baseline up to 48 weeks after completion of study treatment
  Patients will be evaluated using the 6 minute walk test, single leg stance, and functional reach and grip strength using a dynamometer.
Change in ability to perform routine activities | Baseline up to 48 weeks after completion of study treatment
  Patients will be evaluated using the human activity profile and activity card sort.
Change in pain | Baseline up to 48 weeks after completion of study treatment
  Patients will be evaluated using the comparative pain scale.
Change in fine motor dexterity | Baseline up to 48 weeks after completion of study treatment
  Patients will be evaluated using the the group peg board test.
Change in overall quality of life | Baseline up to 48 weeks after completion of study treatment
  Improvement of patients' overall quality of life will be evidence of response, and assessments will be made at baseline and throughout the trial, as well as at the conclusion of the trial, to evaluate for any improvement in quality of life. Patients will be evaluated using the National Institute of Neurological Disorders and Stroke-Neuro-Quality of Life scale.
Resistance to therapy | Up to 1 year
  Resistance to therapy will be evaluated through imaging studies and patient follow up for at least one year, but this is not expected with the combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm